CLINICAL TRIAL: NCT05962151
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Two-Period Crossover Efficacy and Safety Study of Nalbuphine ER Tablets for the Treatment of Refractory Chronic Cough
Brief Title: Refractory Chronic Cough Improvement Via NAL ER (RIVER)
Acronym: RIVER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trevi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NAL04-201
Record Dates: First submitted 2023-07-07; First posted 2023-07-27 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Refractory Chronic Cough
Keywords: RCC; Cough; Nalbuphine
MeSH Terms: conditions — Chronic Cough; Cough | interventions — Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- First NAL ER, then Placebo (Experimental): Participants will receive NAL ER at escalating doses (27 mg QD to BID, 54 mg BID, and 108 mg BID) in Treatment Period 1, followed by placebo matched to NAL ER in Treatment Period 2.
  Interventions: Drug: NAL ER; Drug: Placebo
- First Placebo then NAL ER (Experimental): Participants will receive placebo matched to NAL ER in Treatment Period 1, followed by NAL ER at escalating doses (27 mg QD to BID, 54 mg BID, and 108 mg BID) in Treatment Period 2.
  Interventions: Drug: NAL ER; Drug: Placebo

INTERVENTIONS:
Drug: NAL ER — Oral tablets
  Other Names: Nalbuphine
Drug: Placebo — Oral tablets

SUMMARY:
The main purpose of this study is to evaluate the effect of NAL ER on 24-hour cough frequency and to assess safety and tolerability of NAL-ER for treatment of refractory chronic cough.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of refractory chronic cough (RCC) for at least one year
* Chest radiograph or CT of thorax within 24 months or during screening not demonstrating any significant abnormalities contributing to RCC

Exclusion Criteria:

* Diagnosis of sleep apnea
* Respiratory tract infection within 6 weeks of Baseline
* History of bronchiectasis, COPD, or IPF
* History of uncontrolled asthma
* Current smokers/vapers, quit smoking with <=12 months, using nicotine supplements, or history of >=20 pack years
* History of major psychiatric disorder
* History of substance abuse
* Pregnant or lactating females
* Known intolerance to opioids
* Abnormal kidney or liver functions based on Screening lab results.
* Known hypersensitivity to nalbuphine or to NAL ER excipients
* Previous participation in a nalbuphine ER clinical study
* Use of opiates, benzodiazepines, or MAOIs within 14 days of Baseline
* Use of pregabalin, gabapentin, thalidomide for treatment of cough within 14 days of Baseline
* Use of ACE inhibitors within 12 weeks of Baseline
* Use of a medication having a "known risk" of Torsade de Pointes (categorized as "KR" on the Credible Meds® website.) 4 weeks prior to Baseline
* Use of unstable doses of medications associated with a potential risk of QT prolongation but not clearly associated with Torsade de Pointes within 4 weeks of screening.
* Use of unstable doses of cough suppressants within 14 days of Baseline
* Use of unstable doses of medications that affect serotonergic neurotransmission that may cause serotonin syndrome with opioids within14 days of Baseline
* Use of unstable doses of P450 isozyme inhibitors/inducers within 14 days of Baseline

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Relative Change From Baseline in 24-hour Cough Frequency at Day 21 | Baseline, Day 21

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to Week 15
Relative Change From Baseline in 24-hour Cough Frequency at Days 7 and 14 | Baseline, Day 7 and 14
Percentage of Participants With >=30%, 50% and 75% Reduction in 24-hour Cough Frequency at Days 7, 14, and 21 | At Days 7, 14, and 21
Relative Change From Baseline in Awake Cough Frequency at Days 7, 14, and 21 | Baseline, Day 7, 14 and 21
Relative Change From Baseline in Sleep Cough Frequency at Days 7, 14, and 21 | Baseline, Day 7, 14 and 21
Change From Baseline in Cough Severity Visual Analogue Scale at Days 7, 14, and 21 | Baseline, Day 7, 14 and 21
Change From Baseline in Leicester Cough Questionnaire (LCQ) Total Score at Day 21 | Baseline, Day 21
Change From Baseline in Patient-Reported Cough Frequency (PR-CF) at Days 7, 14, and 21 | Baseline, Day 7, 14 and 21
Percentage of PR-CF Responders With at Least one Category Improvement at Days 7, 14, and 21 | At Days 7, 14, and 21
Change From Baseline in Patient Global Impression of Severity (PGI-S) Cough at Days 7, 14, and 21 | Baseline, Day 7, 14 and 21
Absolute Values of Patient Global Impression of Change for Cough (PGI-C) Score at Days 7, 14, and 21 | At Days 7, 14, and 21
Change From Baseline in Clinicians Global Impression of Cough Severity Score at Day 21 | Baseline, Day 21
Absolute Values of Clinicians Global Impression of Change for Cough Score at Day 21 | At Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Trevi Therapeutics
Locations (14):
- Canada (3):
  - McMaster University Medical Centre, Hamilton, Ontario
  - Inspiration Research, Toronto, Ontario
  - CIC Mauricie Inc., Trois-Rivières, Quebec
- United Kingdom (11):
  - Hull and East Yorkshire Hospitals NHS Trust - Castle Hill Hospital, Cottingham, East Riding Of Yorkshire
  - Kings College Hospital NHS Foundation Trust, London, Greater London
  - University Hospital of South Manchester NHS Foundation Trust (UHSM) - Wythenshawe Hospital, Manchester, Greater Manchester
  - Accellacare South London, Orpington, Kent
  - Accellacare North London, Northwood, Middlesex
  - Belfast City Hospital, Belfast, Northern Ireland
  - North Tyneside General Hospital - Northumbria Healthcare NHS Foundation Trust, North Shields, Tynemouth
  - Accellacare Warwickshire, Coventry, Warwickshire
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - Accellacare Yorkshire, Shipley, Yorkshire
  - Egin Research Ltd, High Wycombe

IPD SHARING:
Plan to Share IPD: No